CLINICAL TRIAL: NCT05334641
Title: The Effect of Music on Pain and Anxiety in Patients Receiving Chemotherapy During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulsum Yetis Koca, Lecturer, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: InonuGYKoca001
Record Dates: First submitted 2022-04-17; First posted 2022-04-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cancer; Chemotherapy
Keywords: Anxiety; COVID-19; Music; Pain; Patients receiving chemotherapy
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; COVID-19; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Listening Music
- Control Group (Active Comparator)
  Interventions: Other: Not Listening Music

INTERVENTIONS:
Other: Listening Music — The patients in the experimental group were listened to music.
  Arms: Experimental Group
Other: Not Listening Music — The control group was not listened to music.
  Arms: Control Group

SUMMARY:
Introduction: This study has been conducted to determine the effect of music on pain and anxiety levels in patients receiving chemotherapy during COVID-19.

Methods: The research has been carried out in a real trial model with adult patients receiving chemotherapy. The sample of the study is consisted of 92 patients (45 in the experimental group and 47 for the control group). The data have been collected by the researcher with Google Forms (using State and Transient Anxiety Inventory and Visual Analog Skala) between March 2020 and July 2020, through the links sent to the phones of participants on the day they received chemotherapy.

Results: The mean scores obtained from the post-test STAI (53.11±4.77) and VAS (3.44±2.53) scales in the experimental group have been determined to statistically significantly decrease when compared to the pre-test measurement data (STAI:54.26±4.26; VAS:4.22±2.41) (p<0.05). No statistically significant difference has been determined between pre-test and post-test mean scores of the patients in the control group.

Conclusion: It has been observed that music applications reduce the pain and anxiety levels of patients receiving chemotherapy during the COVID-19 process. It can be recommended to use music applications in the management of pain and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Over the age 18,
* Being able to communicate,
* Being literate,
* Having no diagnosis of psychiatric,
* Have the necessary technological equipment (phone, internet, etc.)

Exclusion Criteria:

* Existing infection
* Receiving palliative chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Google Forms (using State and Transient Anxiety Inventory and Visual Analog Skala) | The posttest was administered 1 hour after the pretest.
  The data have been collected by the researcher with Google Forms (using State and Transient Anxiety Inventory and Visual Analog Skala).The posttest was administered 1 hour after the pretest.

CONTACTS AND LOCATIONS:
Overall Officials: Rukuye AYLAZ, Study Director — Inonu University
Locations (1):
- Vocational School of Health Services, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No